CLINICAL TRIAL: NCT00589797
Title: Clinical Study to Evaluate the Safety and Effectiveness of the Aesculap Activ-L™ Artificial Disc in the Treatment of Degenerative Disc Disease
Brief Title: Activ-L™ Artificial Disc Treatment of Degenerative Disc Disease in the Treatment of Degenerative Disc Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aesculap Implant Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASC-01
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-11

CONDITIONS: Degenerative Disc Disease
Keywords: Degenerative; Disc
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational (Experimental): Implantation of the Activ-L Artificial Disc at one level of the lumbar spine, either L4/L5 or L5/S1.
  Interventions: Device: Activ-L Artificial Disc
- Control (Active Comparator): Implantation of either the ProDisc-L Total Disc Replacement or Charité Artificial Disc at one level of the lumbar spine, either L4/L5 or L5/S1.
  Interventions: Device: ProDisc-L Total Disc Replacement or Charité Artificial Disc

INTERVENTIONS:
Device: Activ-L Artificial Disc — Implantation at one level of the lumbar spine, either L4/L5 or L5/S1.
  Arms: Investigational
Device: ProDisc-L Total Disc Replacement or Charité Artificial Disc — Implantation at one level of the lumbar spine, either L4/L5 or L5/S1.
  Arms: Control

SUMMARY:
The purpose of this study is to learn whether an investigational device called the Activ-L Artificial Disc is safe and effective in the treatment of degenerative disc disease of the lower (lumbar) spine.

DETAILED DESCRIPTION:
The objective of this clinical study is to evaluate the safety and effectiveness of the Activ-L Artificial Disc for treatment of single-level degenerative disc disease of the lumbar spine in patients who have been unresponsive to at least six months of prior conservative care. The hypothesis of the study is that the Activ-L Disc is non-inferior to the control (the Charité® Artificial Disc [DePuy Spine] or ProDisc-L® Total Disc Replacement [Synthes Spine]) with respect to the rate of individual subject success at 24 months. Individual subject success is a composite of effectiveness and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 60, skeletally mature
* Symptomatic DDD with objective evidence of lumbar DDD, with any of the following characteristics by MRI scan:

  * instability as defined by ≥ 3mm translation or ≥ 5° angulation.
  * osteophyte formation of facet joints or vertebral endplates.
  * decreased disc height of >2mm as compared to the adjacent level.
  * scarring/thickening of the ligamentum flavum, annulus fibrosis, or facet joint capsule.
  * herniated nucleus pulposus.
  * facet joint degeneration/changes.
  * vacuum phenomenon.
* Single level symptomatic disease at L4/L5 or L5/S1.

  * six months of unsuccessful conservative treatment
* ODI score ≥ 40/100.
* Surgical candidate for an anterior approach to the lumbar spine.
* Back pain at the operative level only, with or without leg pain.
* Back pain VAS score greater than the higher of the two VAS leg pain scores.
* VAS back pain score ≥ 40/100 mm.
* Willing to return for follow-up visits and sign an Informed Consent and HIPAA Authorization.

Exclusion Criteria:

* Previous surgery at any lumbar level, except IDET (Intradiscal Electrothermal Annuloplasty), percutaneous nucleoplasty, or microdiscectomy.
* Chronic radiculopathy, i.e., subject complaint of unremitting pain with a predominance of leg pain symptoms greater than back pain symptoms extending over a period of at least 1 year.
* endplate dimensions smaller than 34.5 mm in medial-lateral and/or 27 mm in the anterior-posterior direction
* Evidence of significant, symptomatic disc degeneration at another lumbar level.
* Preoperative remaining disc height < 3mm
* Myelopathy.
* Previous compression or burst fracture at the affected level.
* Sequestered herniated nucleus pulposus with migration.
* Mid-sagittal stenosis of <8mm (by MRI).
* Degenerative or lytic spondylolisthesis > 3mm.
* Spondylolysis.
* Isthmic spondylolisthesis.
* Lumbar scoliosis (> 11 degrees of sagittal plane deformity).
* Spinal tumor.
* Active systemic infection or infection at the site of surgery.
* Facet ankylosis or severe facet degeneration.
* Continuing steroid use or prior use for more than 2 months.
* History of allergies to any of the device components.
* Pregnancy or planning to become pregnant within the next 2 years.
* Morbid obesity (BMI >35).
* Investigational drug or device use within 30 days.
* Osteoporosis or osteopenia
* Metabolic bone disease.
* Leg pain with migrated sequestrum fragment.
* History of rheumatoid arthritis, lupus, or other autoimmune disorder.
* Ankylosing spondylitis.
* History of HIV/AIDS or hepatitis that precludes surgery.
* History of deep vein thrombosis, symptoms of arterial insufficiency, or thromboembolytic disease.
* Current or recent history of illicit drug or alcohol abuse, or dependence as defined as the continued use of alcohol despite the development of social, legal, or health problems.
* Life expectancy <5 years.
* Chemotherapy within past 5 years or any cancer other than non-melanoma skin cancer treated with curative intent within the past 5 years.
* Prior nephrectomy.
* Abdominal adhesions, endometriosis, inflammatory bowel disease, Crohn's disease, diverticulitis, ulcerative colitis or other abdominal pathology that would preclude abdominal surgical approach.
* Insulin-dependent diabetes.
* Any degenerative muscular or neurological condition that would interfere with evaluation of outcomes, including but not limited to Parkinson's disease, ALS (amyotrophic lateral sclerosis), or multiple sclerosis.
* History of Pelvic Inflammatory Disease.
* Peritonitis.
* Currently in active spinal litigation as a result of medical negligence.
* Prisoner.
* Psychiatric or cognitive impairment that would interfere with the subject's ability to comply with the study requirements, e.g., Alzheimer's disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 376 (Actual)
Dates: Start 2007-01; Primary Completion 2012-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolando Garcia, M.D., Principal Investigator — Orthopedic Care Center; James J Yue, M.D., Principal Investigator — Yale University; Dom Coric, M.D., Principal Investigator — Carolina Neurosurgery and Spine Associates; Steven Dennis, M.D., Principal Investigator — Hoag Memorial Hospital Presbyterian; Federico P. Girardi, M.D., Principal Investigator — Hospital for Special Surgery, New York; Mick Perez-Cruet, M.D., Principal Investigator — Michigan Head and Spine Institute; Harel Deutsch, M.D., Principal Investigator — Rush University Medical Center; Glenn Buttermann, M.D., Principal Investigator — Midwest Spine Institute; Dzung Dinh, M.D., Principal Investigator — Neuroscience Education and Research Foundation; Vikas Patel, M.D., Principal Investigator — University of Colorado, Denver; Christopher Ames, M.D., Principal Investigator — University of California, San Francisco; John Regan, M.D., Principal Investigator — St. John's Hospital and Health Center; Andrew Dailey, M.D., Principal Investigator — University of Utah Medical Center; Darren Bergey, M.D., Principal Investigator — Rancho Specialty Hospital; Brian Dalton, M.D., Principal Investigator — Hamot Medical Center; Scott Leary, M.D., Principal Investigator — Scripps Memorial Hospital La Jolla; David Hart, M.D., Principal Investigator — University Hospitals Cleveland; Antonio Castellvi, M.D., Principal Investigator — Foundatin for Orthopaedic Research and Education
Locations (17):
- United States (17):
  - Scripps Memorial Hospital La Jolla, La Jolla, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Rancho Specialty Hospital, Rancho Cucamonga, California
  - University of California San Francisco, San Francisco, California
  - St. John's Hospital and Health Center, Santa Monica, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Yale University School of Medicine/New Haven Hospital, New Haven, Connecticut
  - Aventura Hospital and Medical Center, Aventura, Florida
  - University Community Hospital, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Neurosciences Education and Research Foundation, Peoria, Illinois
  - HealthEast St. John's Hospital, Maplewood, Minnesota
  - Hospital for Special Surgery, New York, New York
  - Carolinas Healthcare, Charlotte, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Hamot Medical Center, Erie, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yue JJ, Mo FF. Clinical study to evaluate the safety and effectiveness of the Aesculap Activ-L artificial disc in the treatment of degenerative disc disease. BMC Surg. 2010 Apr 9;10:14. doi: 10.1186/1471-2482-10-14. PMID 20380708

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 19 US health care center sites
Groups:
- Control: Implantation of either the ProDisc Total Disc Replacement or the Charité Artificial Disc at one level of the lumbar spine, either L4/L5 or L5/S1.
Period: Overall Study
Arm/Group | Investigational | Control
Started | 264 | 112
Baseline | 218 | 106
24 Months | 191 | 89
Completed | 191 | 89
Not Completed | 73 | 23
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 12 | 9
Not completed — Physician Decision | 8 | 3
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Non-Randomized Training Subjects | 46 | 6

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational | Control | Total
Number analyzed (Participants) | 264 | 112 | 376
Age, Categorical [Count of Participants; unit: Participants] — All enrolled subjects
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 264 | 112 | 376
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — All enrolled subjects
  years | 39.1 (8.6) | 40.0 (8.6) | 39.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants] — All enrolled subjects
  Participants
    Female | 124 | 56 | 180
    Male | 140 | 56 | 196
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — All enrolled subjects
  Participants
    Hispanic or Latino | 29 | 12 | 41
    Not Hispanic or Latino | 235 | 100 | 335
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — All enrolled subjects
  Participants
    American Indian or Alaska Native | 3 | 0 | 3
    Asian | 3 | 0 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 18 | 5 | 23
    White | 233 | 106 | 339
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 7 | 1 | 8
Oswestry Disability Index (ODI) Scores for Low Back Pain [Mean (Standard Deviation); unit: units on a scale] — Scores on a scale from 0 (minimal disability) to 100 (bed-bound)
  units on a scale | 57.1 (13.9) | 58.6 (14.1) | 57.9 (13.9)
Visual Analog Scale (VAS) Ratings for Back and Leg Pain [Mean (Standard Deviation); unit: units on a scale] — Ratings on a scale from 0 (no pain) to 100 (worst possible pain)
  units on a scale
    VAS Back Pain | 79.0 (14.9) | 79.1 (14.8) | 79.1 (14.8)
    VAS Right Leg Pain | 28.7 (29.8) | 32.9 (29.6) | 30.6 (30.0)
    VAS Left Leg Pain | 29.6 (29.4) | 30.7 (29.5) | 30.4 (29.6)
Short-Form (36) Health Questionnaire (SF-36) Scores [Mean (Standard Deviation); unit: units on a scale] — Scores on a scale from 0 (maximum disability) to 100 (no disability) for mental component summary (MCS) and physical component summary (PCS)
  units on a scale
    SF-36 MCS | 39.1 (13.9) | 39.6 (14.9) | 39.4 (14.4)
    SF-36 PCS | 29.9 (6.2) | 28.4 (6.2) | 29.2 (6.2)
Rotational Range of Motion [Mean (Standard Deviation); unit: degrees]
  Flexion/Extension | 6.6 (5.1) | 6.6 (4.6) | 6.6 (4.8)
  Lateral Bending AP | 1.0 (2.0) | 1.0 (1.8) | 1.0 (1.9)
Translational Range of Motion [Mean (Standard Deviation); unit: millimeters] | 0.5 (0.7) | 0.6 (0.6) | 0.6 (0.6)
Normal Neurological Status [Number; unit: participants] — Number of subjects meeting the following criteria for normal status: Motor - Grade 5 (active movement vs. full resistance); Sensory - Grade 2 (normal); Reflexes - Grade 2 (normal)
  participants
    Motor | 97 | 40 | 137
    Sensory | 78 | 33 | 111
    Reflexes | 91 | 42 | 133

OUTCOME MEASURES:

1. Primary Outcome: Overall Success at 24 Months Relative to Baseline
Description: Measured by absence of treatment failure; absence or serious device related AE; maintenance or improvement of ROM at index level; maintenance or improvement of neurological status; improvement in ODI score.
Time Frame: 24 months
Population: Intent to treat population; missing data imputed as failures
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 218 | 106
percentage of participants
  Including ROM success component | 42.2 [35.6 to 49.1] | 28.3 [20.0 to 37.9]
  Without ROM success component | 61.9 [55.1 to 68.4] | 52.8 [42.9 to 62.6]
Statistical Analysis 1: Comparison: Investigational vs Control; Test type: Non-Inferiority — The trial was designed as a non-inferiority trial with a margin (delta) of 15%. Additional analyses using a delta of 10% as requested by FDA were also conducted; p < 0.05, t-test, 1 sided

2. Secondary Outcome: VAS Success for Back and Leg Pain at Rest
Description: Number of patients demonstrating improvement in back and leg pain at 24 months compared to baseline
Time Frame: 24 months
Population: Intent to treat population; observed data (i.e. missing data not imputed as failures)
Measure: Number; unit: participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 180 | 84
participants
  VAS Rating for Back Pain | 162 | 72
  VAS Rating for Left Leg Pain | 72 | 35
  VAS Rating for Right Leg Pain | 73 | 36

3. Primary Outcome: Device Success
Description: Percent of subjects demonstrating no Subsequent Surgical Interventions (SSI's) at the index level (L4-L5 or L5-S1) at 24 months.
Time Frame: 24 months
Population: Intent to treat population; missing data imputed as failures
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 218 | 106
percentage of participants | 84.4 [78.9 to 89.0] | 84.9 [76.6 to 91.1]

4. Primary Outcome: Absence of Serious Device Related Adverse Events
Description: Percent of subjects demonstrating no device related SAE's at 24 months as per the Clinical Events Committee (CEC)
Time Frame: 24 months
Population: Intent to treat population; missing data imputed as failures
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 218 | 106
percentage of participants | 76.6 [70.4 to 82.1] | 70.8 [61.1 to 79.2]

5. Primary Outcome: Range of Motion (ROM) Success
Description: Percent of subjects demonstrating maintenance or improvement in ROM at 24 months compared to baseline
Time Frame: 24 months
Population: Intent to treat population; missing data imputed as failures
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 218 | 106
percentage of participants | 58.7 [51.9 to 65.3] | 42.5 [32.9 to 52.4]

6. Primary Outcome: Neurological Success
Description: Percent of patients demonstrating maintenance or improvement in combined motor and sensory evaluations at 24 months compared to baseline
Time Frame: 24 months
Population: Intent to treat population; missing data imputed as failures
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 218 | 106
percentage of participants | 80.3 [74.4 to 85.3] | 76.4 [67.2 to 84.1]

7. Primary Outcome: ODI Success
Description: Percent of subjects demonstrating an improvement of greater than or equal to 15 points at 24 months compared to baseline
Time Frame: 24 months
Population: Intent to treat population; missing data imputed as failures
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 218 | 106
percentage of participants | 75.2 [68.9 to 80.8] | 66.0 [56.2 to 75.0]

8. Secondary Outcome: ODI Success Using Two Measures of Success
Description: Number of subjects demonstrating improvement in two measures of ODI success at 24 months compared to baseline
Time Frame: 24 months
Population: Intent to treat population; observational data (i.e. missing data not imputed as failures)
Measure: Number; unit: participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 187 | 87
participants
  Greater than or equal to 15 points of improvement | 164 | 70
  Greater than or equal to 15% improvement | 170 | 77

9. Secondary Outcome: Improvement in SF-36 Scores
Description: Number of subjects demonstrating a greater than or equal to 15% improvement in mental (MCS) and physical (PCS) component summary scores at 24 months compared to baseline
Time Frame: 24 months
Population: Intent to treat population; observational data (i.e. missing data not imputed as failures)
Measure: Number; unit: participants
Arm/Group | Investigational | Control
Number analyzed (Participants) | 180 | 86
participants
  SF-36 MCS | 101 | 48
  SF-36 PCS | 156 | 69

ADVERSE EVENTS:
Time Frame: Serious and Non-Serious Adverse Events Adjudicated as of 9 October 2015
Description: All anticipated and unanticipated serious and non-serious adverse events in the intent to treat population
Arm/Group | Investigational | Control
Serious Adverse Events (participants affected / at risk) | 86/218 | 57/106
Other Adverse Events (participants affected / at risk) | 197/218 | 100/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational (N=218) | Control (N=106)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
High Cholesterol (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac Issues (Cardiac disorders) | 5 (5) | 0 (0) — Includes arrhythmia, chest pain, heart disease and myocardial infarct
Eyes, Ears, Nose or Throat Issues (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Diabetes Mellitus (Endocrine disorders) | 4 (4) | 1 (1)
Goiter (Endocrine disorders) | 1 (1) | 0 (0)
Esophageal Issues (Gastrointestinal disorders) | 1 (1) | 1 (1) — Includes esophageal bleeding and esophagitis
Gastric Issues (Gastrointestinal disorders) | 3 (3) | 2 (2) — Includes abdominal pain, stomach flu, gastric infection and peptic ulcer
Intestinal Issues (Gastrointestinal disorders) | 5 (5) | 5 (5) — Includes appendicitis and bowel obstruction
Other GI Issues (Gastrointestinal disorders) | 4 (4) | 0 (0) — Includes weight gain, colonoscopy and hernia repair
Gall Bladder Issues (Hepatobiliary disorders) | 4 (4) | 3 (3) — Includes cholecystectomy, cholecystitis and gallstones
Liver Fibrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Fever (Immune system disorders) | 1 (1) | 0 (0)
Sjogren's Syndrome (Immune system disorders) | 0 (0) | 1 (1)
Systemic Allergic Reaction (Immune system disorders) | 1 (1) | 1 (1)
Systemic Infection (Infections and infestations) | 1 (1) | 1 (1)
Trauma (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) — Includes motor vehicle accident, fall, trip, slip or twist
Bone Fracture - Lumbar (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone Fracture - Non-Lumbar (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Degenerative Joint Disease - Lumbar (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) — Includes arthritis, facet joint degeneration and rheumatoid arthritis
Degenerative Joint Disease - Non-Lumbar (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Includes inflammatory polyarthritis
Joint or Muscle Issues (Musculoskeletal and connective tissue disorders) | 10 (11) | 0 (0) — Includes ganglion cyst, hallux rigidus, hip-joint pain, surgery, torn meniscus and trigger finger
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Non-Lumbar Radiographic Observation (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) — Includes disc bulge and disc herniation
Pain in Non-Lumbar or Leg (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) — Includes neck and thoracic
Plantar Fascitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (14) | 5 (5) — Includes breast, colon, prostate, rectal, skin and vulvar
Lower Extremity Pain (Nervous system disorders) | 7 (7) | 4 (4) — Includes bilateral lower leg, unilateral upper and lower leg
Lumbar Only Pain (Nervous system disorders) | 6 (6) | 6 (6)
Lumbar and Lower Extremeties Sensory Deficit (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar and Lower Extremities Motor Deficit (Nervous system disorders) | 2 (2) | 0 (0) — Includes general and transient unilateral motor deficit
Lumbar and Lower Extremity Pain (Nervous system disorders) | 9 (9) | 8 (8) — Includes lumbar + unilateral and bilateral radiation into upper and lower leg
Non-Lumbar and Lower Extremities Deficit (Nervous system disorders) | 3 (3) | 4 (4) — Includes brain tumor, headache, loss of consciousness, nerve entrapment, seizure, vertigo and carpal tunnel syndrome
Pregnancy Related Issues (Pregnancy, puerperium and perinatal conditions) | 7 (8) | 1 (1) — Includes pregnancy, delivery and miscarriages
Psychosocial Disorders (Psychiatric disorders) | 1 (1) | 3 (3) — Includes conversion disorder, depression and suicidal attempt
Substance Related Disorders (Psychiatric disorders) | 4 (4) | 2 (2) — Includes substance dependence and withdrawal
Suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Benign Prostatic Hypertrophy (Renal and urinary disorders) | 1 (1) | 0 (0)
Kidney Issues (Renal and urinary disorders) | 2 (2) | 1 (1) — Includes kidney stones
Female Reproductive System Issues (Reproductive system and breast disorders) | 3 (3) | 2 (2) — Includes breast implant leakage, irregular menstrual bleeding and ovarian or uterine cyst or mass or tumor
Male Reproductive System Issues (Reproductive system and breast disorders) | 5 (5) | 4 (4) — Includes erectile dysfunction and retrograde ejaculation
Reproductive System Related Surgeries (Reproductive system and breast disorders) | 3 (3) | 1 (1) — Includes breast reduction or enhancement and hysterectomy
Breathing Disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Includes dyspnea
Respiratory Infections (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) — Includes bronchitis and pneumonia
Device Deficiency (Surgical and medical procedures) | 7 (7) | 3 (3) — Includes implant expulsion, malposition, migration and subsidence
Index Procedure Related Wounds (Surgical and medical procedures) | 4 (4) | 2 (2) — Includes deep wounds, dural injuries and incisional hernia
Subsequent Surgical Intervention Procedure Related Wounds (Surgical and medical procedures) | 0 (0) | 1 (1) — Includes incisional hernia
Blood Loss (Vascular disorders) | 1 (1) | 0 (0)
Blood Pressure (Vascular disorders) | 1 (1) | 2 (2) — Includes syncope
Embolism (Vascular disorders) | 1 (1) | 0 (0) — Includes pulmonary embolism
Thrombosis (Vascular disorders) | 2 (2) | 0 (0) — Includes deep vein thrombosis
Vascular Issues (Vascular disorders) | 1 (1) | 3 (3) — Includes aneurysm, atherosclerosis and iliac vessel tear
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational (N=218) | Control (N=106)
Blood Pressure (Vascular disorders) | 9 (9) | 7 (7) — Includes hypertension and syncope
Vascular Issues (Vascular disorders) | 4 (4) | 1 (1) — Includes aneurysm, arterial dissection, atherosclerosis and iliac vessel tear
Cardiac Issues (Cardiac disorders) | 4 (4) | 3 (3) — Includes arrhythmia, chest pain, heart disease and myocardial infarct
Diabetes Mellitus (Endocrine disorders) | 4 (4) | 0 (0)
Eyes, Ears, Nose or Throat (Ear and labyrinth disorders) | 6 (6) | 6 (6)
Gastric Issues (Gastrointestinal disorders) | 27 (27) | 9 (10) — Includes abdominal adhesion, abdominal pain, acid reflux, indigestion, food poisoning, GERD, gastric lesions, gastritis, stomach flu, gastrointestinal infection and peptic ulcer
Intestinal Issues (Gastrointestinal disorders) | 16 (17) | 11 (13) — Includes bowel irregularity, constipation, diverticulitis, GI bleed, inflammatory bowel syndrome, nausea, vomiting and diarrhea
Pregnancy Related Issues (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3) — Includes pregnancy and delivery
Male Reproductive System Issues (Reproductive system and breast disorders) | 7 (8) | 3 (3) — Includes epididymitis, erectile dysfunction, inguinal or testicular pain, rectocele and retrograde ejaculation
Female Reproductive System Issues (Reproductive system and breast disorders) | 6 (6) | 1 (1) — Includes abnormal PAP smear results, breast, ovarian or uterine cyst, mass or tumor, cystocele, menopause, vaginal or yeast infection
Reproductive System Related Surgeries (Reproductive system and breast disorders) | 4 (4) | 0 (0) — Includes abortion, hysterectomy and lumpectomy
Urinary Issues (Renal and urinary disorders) | 23 (24) | 7 (8) — Includes decreased urine output, bladder infection, hematuria, incontinence, dysuria, pelvic pain, urinary hesitance, retention, urgency or tract infection
Non-Procedure Allergic Reactions (Immune system disorders) | 3 (3) | 5 (5) — Includes seasonal and systemic allergic reactions
Infections (Infections and infestations) | 4 (4) | 2 (2) — Includes abscess, cellulitis and non-procedure wound infections
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
High Cholesterol (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
Degenerative Joint Disease - Lumbar (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) — Includes ankylosing spondylitis, arthritis, arthropathy and facet joint degeneration
Plantar Fascitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Joint or Muscle Issues (Musculoskeletal and connective tissue disorders) | 19 (22) | 11 (13) — Includes non-lumbar benign mass or tumor, bursitis, ganglion cyst, gout, hallux rigidus, hiccups, hip joint pain, non-lumbar joint sprain, leg length discrepancy, SI joint pain, surgery, torn meniscus, torn hip labral tear and trigger finger
Pain in Non-Lumbar or Leg (Musculoskeletal and connective tissue disorders) | 45 (54) | 14 (15) — Includes ankle, back, upper extremities, neck and thoracic, fibromyalgia, and foot
Non-Lumbar Radiographic Observation (Surgical and medical procedures) | 19 (19) | 9 (9) — Includes disc bulge, protrusion and herniation
Lumbar and Lower Extremity Motor Deficit (Musculoskeletal and connective tissue disorders) | 6 (7) | 5 (6) — Includes general, persistent and transient unilateral and bilateral motor deficit
Lumbar and Lower Extremity Sensory Deficit (Musculoskeletal and connective tissue disorders) | 24 (25) | 16 (18) — Includes unilateral and bilateral general and upper extremity sensory deficit, positive or change in SLR test
Reflex Change or Abnormality (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1)
Non-Lumbar and Lower Extremity Deficit (Nervous system disorders) | 18 (19) | 7 (8) — Includes Bell's palsy, brain tumor, dysphagia, memory loss, headache, loss of consciousness, migraine, nerve entrapment, numbness, restlessness, seizure, tremor, vertigo, carpal tunnel, peripheral neuropathy, upper extremity motor/sensory deficits
Lower Extremity Pain (Nervous system disorders) | 40 (45) | 11 (15) — Includes unilateral and bilateral upper and lower leg
Lumbar Only Pain (Nervous system disorders) | 44 (48) | 30 (31)
Lumbar and Lower Extremity Pain (Nervous system disorders) | 42 (42) | 23 (23) — Includes lumbar + unilateral and bilateral radiation into upper and lower leg
Psychosocial Disorders (Psychiatric disorders) | 12 (15) | 5 (5) — Includes anxiety, bipolar and depressive disorders
Substance Related Disorders (Psychiatric disorders) | 6 (6) | 1 (1) — Includes substance dependence or withdrawal
Sleep Disorders (Psychiatric disorders) | 6 (6) | 2 (2) — Includes fatigue, sleepiness, somnolence and insomnia
Breathing Disorders (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) — Includes dyspnea, sleep apnea, cough and asthma
Respiratory Infections (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6) — Includes bronchitis, respiratory and sinus infection
Other Respiratory Disorders (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) — Includes COPD, hemoptysis, pleuritic chest pain, reactive airway disease
Trauma (Injury, poisoning and procedural complications) | 38 (50) | 21 (27) — Includes motor vehicle accident, fall, trip, slip or twist
Index Procedure Related Wounds (Surgical and medical procedures) | 17 (18) | 12 (12) — Includes abscess, deep wound, dehiscence, dural injuries, erythema, drainage, inflammation, incisional hernia, incisional cellulitis, pain at incision site, suture reaction and wound infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days